CLINICAL TRIAL: NCT01875159
Title: Pilot Study of Effects of Caffeine on Intermittent Hypoxia in Infants Born Preterm
Brief Title: Effects of Caffeine on Intermittent Hypoxia in Infants Born Preterm
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American SIDS Institute (Other)
Responsible Party: Principal Investigator, Carl Hunt, Research Professor of Pediatrics, American SIDS Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASI 01
Record Dates: First submitted 2013-06-03; First posted 2013-06-11 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Hypoxia
Keywords: Prematurity; Apnea of prematurity; Intermittent hypoxia
MeSH Terms: conditions — Hypoxia; Premature Birth; Apnea | interventions — caffeine citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine (Experimental): Caffeine citrate 6 mg/kg/day
  Interventions: Drug: Caffeine citrate 6 mg/kg/day
- Active Comparator: no caffeine (No Intervention): Compare extended use of caffeine citrate 6 mg/kg/day to no caffeine (usual care) in regard to extent of intermittent hypoxia from 35 weeks postmenstrual age (PMA) to 40 weeks PMA.

INTERVENTIONS:
Drug: Caffeine citrate 6 mg/kg/day — Comparison of caffeine citrate 6 mg/kg/day versus no caffeine (usual care) on extent of intermittent hypoxia at 35, 36, 37, 38, 39, and 40 weeks postmenstrual age.
  Other Names: Cafcit
  Arms: Caffeine

SUMMARY:
The purpose of this pilot study is to document the extent to which intermittent hypoxia persists beyond the age of discontinuing clinical methylxanthine, and will assess the effect of caffeine treatment on the number of intermittent hypoxia episodes and the total number of seconds with a hemoglobin oxygen saturation (HbO2 SAT) below 90%.

DETAILED DESCRIPTION:
Infants with prior clinical treatment with caffeine in the neonatal intensive care unit (NICU) will be enrolled and continuous physiologic data recording of oxygen hemoglobin saturation (HbO2 SAT) and heart rate will begin as early as 33 weeks postmenstrual age (PMA). Randomization will occur when enrolled infants reach a corrected gestational age of at least 34 weeks PMA AND clinical caffeine has been discontinued for at least 5 days. Infants will be randomized to receive caffeine or to continue with usual care. The group randomized to start caffeine will receive an oral loading dose of caffeine citrate of 20 mg/kg on Day #1, followed by a single daily oral maintenance dose of 6 mg/kg starting on Day #2 and continued daily thereafter until 40 weeks PMA. The continuous oximeter recordings will be stopped at the same time. The number of intermittent hypoxia events/hour per week will be compared between the caffeine group and the usual care (no-caffeine) group for each week of physiologic data recordings.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age of 25 + 0 to 32 + 0 weeks PMA at birth, and 34 + 0 to 375 + 6 weeks PMA at randomization
2. Prior treatment with caffeine based on routine clinical indications, and clinical caffeine now discontinued ≥5 days before randomization
3. Previously tolerated clinical treatment with caffeine
4. Breathing room air (no current supplemental O2 treatment; may have previously required respiratory support)
5. Parental consent to enroll in pilot study

Exclusion Criteria:

1. Congenital syndrome or other medical diagnosis associated with known risk for neurodevelopmental abnormality, including intraventricular hemorrhage Grade 3 or greater, cyanotic congenital heart disease, confirmed central nervous system infection, or fetal alcohol syndrome
2. Currently receiving supplemental oxygen, ventilatory support, or nasal airflow therapy
3. Clinical decision to restart caffeine prior to completing 5 days of continuous physiologic monitoring after clinical caffeine stopped
4. Anticipated inability to meet protocol requirements

Ages: 33 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betty McEntire, PhD, Study Director — American SIDS Instittute
Locations (1):
- Uniformed Services University of Health Sciences, Bethesda, Maryland, United States

REFERENCES:
- [Result] Rhein LM, Dobson NR, Darnall RA, Corwin MJ, Heeren TC, Poets CF, McEntire BL, Hunt CE; Caffeine Pilot Study Group. Effects of caffeine on intermittent hypoxia in infants born prematurely: a randomized clinical trial. JAMA Pediatr. 2014 Mar;168(3):250-7. doi: 10.1001/jamapediatrics.2013.4371. PMID 24445955

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Caffeine | Active Comparator: no Caffeine
Started | 45 | 53
Completed | 42 | 53
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caffeine | Active Comparator: no Caffeine | Total
Number analyzed (Participants) | 45 | 53 | 98
Age, Customized [Mean (Standard Deviation); unit: Weeks]
  Gestational Age | 28.6 (1.7) | 29.1 (1.7) | 28.9 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 47
  Male | 24 | 27 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 8 | 10
  Not Hispanic or Latino | 40 | 45 | 85
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 11 | 9 | 20
  White | 27 | 42 | 69
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 45 | 53 | 98
Mean birth weight [Mean (Standard Deviation); unit: grams] | 1262.1 (265.6) | 1274.5 (270.3) | 1270.1 (267.2)

OUTCOME MEASURES:

1. Primary Outcome: Episodes of Intermittent Hypoxia Per Hour
Description: Number of episodes of Intermittent hypoxia per hour of pulse oximeter recording less than 90% oxygen saturation
Time Frame: 35, 36, 37, 38 weeks postmenstrual age
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: Events per hour
Arm/Group | Caffeine | Active Comparator: no Caffeine
Number analyzed (Participants) | 42 | 53
Events per hour
  Week 35 | 3.6 (4.3) | 8.4 (8.4)
  Week 36 | 3.8 (4.5) | 8.2 (11.5)
  Week 37 | 4.3 (5.9) | 5.2 (6.8)
  Week 38 | 4.2 (5.7) | 4.7 (6.1)
Statistical Analysis 1: Comparison: Caffeine vs Active Comparator: no Caffeine; >80% probability of detecting at least a 36% reduction in intermittent hypoxia events/hour of recording and in sec/hour <90% oxygen saturation/hour of recording; Test type: Superiority or Other; p < 0.05, GEE gamma regression models

2. Primary Outcome: Number of Seconds of Intermittent Hypoxia Per Hour
Description: Number of seconds of Intermittent hypoxia per hour of pulse oximeter recording less than 90% oxygen saturation
Time Frame: 35, 36, 37, 38 weeks postmenstrual age
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: seconds per hour
Arm/Group | Caffeine | Active Comparator: no Caffeine
Number analyzed (Participants) | 42 | 53
seconds per hour
  Week 35 | 50.9 (48.1) | 106.3 (89.0)
  Week 36 | 49.5 (52.1) | 100.1 (114.6)
  Week 37 | 58.8 (74.1) | 66.8 (75.2)
  Week 38 | 69.3 (108.8) | 66.0 (74.8)

ADVERSE EVENTS:
Arm/Group | Caffeine | Active Comparator: no Caffeine
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/53
Other Adverse Events (participants affected / at risk) | 5/42 | 0/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caffeine (N=42) | Active Comparator: no Caffeine (N=53)
Tachycardia (Cardiac disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No